CLINICAL TRIAL: NCT04328623
Title: Interest of Hypnosis on Pain Management During a Guided Echo Infiltration of the Hand
Acronym: HYMN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Departemental Vendee (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: CHD 202-19
Record Dates: First submitted 2020-03-30; First posted 2020-03-31 (Actual); Results first posted 2024-08-15 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2025-11

CONDITIONS: Hand Injuries
MeSH Terms: conditions — Hand Injuries | interventions — Hypnosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Infiltration (Active Comparator): Ultrasound-guided hand infiltration
  Interventions: Procedure: Infiltration
- Hypnosis (Experimental): Hypnosis before Ultrasound-guided hand infiltration
  Interventions: Procedure: Hypnosis; Procedure: Infiltration

INTERVENTIONS:
Procedure: Hypnosis — conversational hypnosis technique call the "magic glove"
  Arms: Hypnosis
Procedure: Infiltration — Ultrasound-guided hand infiltration

SUMMARY:
Ultrasound-guided infiltration is a common procedure and is known to be locally painful. This care-induced pain leads to strong apprehension in patients who need to benefit from this procedure.

The practice of hypnosis to improve the patient's comfort during a treatment has appeared progressively in hospital departments.

Among the various existing conversational hypnosis techniques, there is the "magic glove" technique. This is the technique that will be used in this study.

The investigators wish to evaluate the interest of hypnosis on the pain felt by the patient when performing an echo-guided infiltration of the hand, one of the most painful extremities during infiltrations.

ELIGIBILITY:
Inclusion Criteria:

* Patient with an indication of a first hand infiltration under ultrasound examination
* Major patient
* Patient with capacity to understand the protocol and has given oral consent to participate in the research,
* Patient with social security coverage.

Exclusion Criteria:

* Patient having preventively applied a pain patch to the area to be infiltrated
* Contraindication to infiltrations ( imbalanced diabetes, imbalanced,hypertension, ongoing infections).
* Hearing impaired patient
* Patient under guardianship/curtel
* Minor
* Pregnant woman
* Patient participating in another intervention research protocol
* Patient unable to follow the protocol as judged by the investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2020-10-08 (Actual); Primary Completion 2022-09-02 (Actual); Study Completion 2022-09-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Adeline Trojet-Bossard, Principal Investigator — CHD Vendée
Locations (1):
- CHD Vendée, La Roche-sur-Yon, France, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Trojet-Bossard A, Dorion A, Planche L, Chollet C, Rabiller S, Cormier G. [Hypnotic pain management during ultrasound-guided infiltration of the hand]. Rev Infirm. 2023 Aug-Sep;72(293):42-44. doi: 10.1016/j.revinf.2023.07.012. Epub 2023 Aug 8. French. PMID 37633694

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Infiltration | Hypnosis
Started | 40 | 40
Infiltration | 40 | 39
Completed | 40 | 39
Not Completed | 0 | 1
Not completed — Protocol Violation | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Infiltration | Hypnosis | Total
Number analyzed (Participants) | 40 | 39 | 79
Age, Continuous [Mean (Standard Deviation); unit: Years] | 60 (11) | 62 (10) | 61 (11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26 | 27 | 53
  Male | 14 | 12 | 26
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Evaluate the Pain Felt in Patients Who Have Benefited From a Hypnosis Session Before a Hand Infiltration Versus Hand Infiltration Without Hypnosis
Description: Analogical visual scale of pain (VAS) To 0mm (no pain) form 10 mm (maximum pain imaginable)
Time Frame: 5 minutes after ultrasound-guided infiltration of hand
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Infiltration | Hypnosis
Number analyzed (Participants) | 40 | 39
units on a scale | 4.56 (2.71) | 1.75 (1.63)
Statistical Analysis 1: Comparison: Infiltration vs Hypnosis; Test type: Superiority; p < 0.001, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: Non applicable
Description: Death, serious adverse events and other (non serious adverse events) were not assessed for the study
Arm/Group | Infiltration | Hypnosis
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-06-14): https://cdn.clinicaltrials.gov/large-docs/23/NCT04328623/Prot_SAP_000.pdf